CLINICAL TRIAL: NCT00459173
Title: Comparison of the Efficacy and Safety of 2 Oral Doses of Rimonabant, 5 mg/Day or 20 mg/Day, Versus Placebo, as an Aid to Maintenance of Smoking Cessation (1-Year Treatment, 1-Year Follow-up)
Brief Title: Efficacy and Safety of Rimonabant as an Aid to Maintenance of Smoking Cessation
Acronym: STRATUS-WW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4796
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2009-04-07 (Estimated); Status verified 2009-04

CONDITIONS: Maintenance of Smoking Cessation
Keywords: abstinence; maintenance
MeSH Terms: interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rimonabant (SR141716)

SUMMARY:
The primary study objective is to evaluate the efficacy of 2 dose levels of rimonabant (5 mg and 20 mg) for the maintenance of abstinence from smoking.

Secondary objectives are to evaluate the effect of rimonabant on craving and weight, the clinical and biological safety of 2 doses of rimonabant rimonabant during a 12-month treatment period and to evaluate the pharmacokinetics of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Smokers smoking at least 10 cigarettes/day as a mean within the 2 months preceding the screening visit
* Motivated to quit with a score greater than or equal to 6 on the ten-point Motivation Scale

Exclusion Criteria:

* non tobacco cigarettes consumption
* chronic use of marijuana
* pregnancy, breastfeeding
* any clinically significant disease that might interfere with the efficacy or safety evaluation of the study drug
* Concomitant use of drugs as an aid to smoking cessation or that might induce weight change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4850 (Actual)
Dates: Start 2002-11; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Time to smoking relapse from the point of re-randomization (Week 10) through Week 32
Smoking relapse defined as: any 7 or more consecutive days of smoking (even a puff) or any 2 consecutive days of smoking 5 or more cigarettes per day

SECONDARY OUTCOMES:
Efficacy: Time to smoking relapse from Week 10 to Week 52, craving, body weight change in abstainers, lipid parameters
Safety data

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Cove, New South Wales, Australia
- Sanofi-Aventis, Laval, Quebec, Canada